CLINICAL TRIAL: NCT06874309
Title: Non-invasive Brain Stimulation to Prepare the Patient for Bariatric Surgery
Brief Title: Non-invasive Brain Stimulation to Prepare the Patient for Bariatric Surgery (REBAS)
Acronym: REBAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Collaborators: St. Anne´s University Hospital Brno (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NW24-04-00392
Record Dates: First submitted 2024-12-19; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: bariatric surgery; obesity; brain stimulation; tDCS; cognitive control; impulsivity; eating behavior
MeSH Terms: conditions — Obesity; Impulsive Behavior; Feeding Behavior | interventions — Bariatric Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active tDCS stimulation (Experimental): Participants in this arm will be stimulated for 4 weeks during weekdays leading to 20 sessions of tDCS over lDLPFC.
  Interventions: Device: home-based tDCS stimulation; Procedure: Bariatric surgery
- sham tDCS stimulation (Sham Comparator): In this arm, sham stimulation will be applied for 4 weeks during weekdays leading to 20 sessions of tDCS over lDLPFC.
  Interventions: Device: home-based tDCS stimulation - sham; Procedure: Bariatric surgery

INTERVENTIONS:
Device: home-based tDCS stimulation — stimulation parameters: 20 sessions of tDCS over lDLPFC (anode over F3, based on the 10:20 system, and cathode over the right supraorbital area), 2 mA intensity, 20 min duration (30 s fade in/fade out)
  Arms: active tDCS stimulation
Device: home-based tDCS stimulation - sham — 20 sessions of tDCS over lDLPFC (anode over F3, based on the 10:20 system, and cathode over the right supraorbital area), the electric current will flow for only 15 s, with similar fade in/fade out, at the beginning and at the end of 20 min, to mimic the subjective sensations that occur during active tDCS.
  Arms: sham tDCS stimulation
Procedure: Bariatric surgery — The operation itself is not a study-related procedure and thus the indicated patients would undergo the surgery regardless of their participation in this study. The operating surgeons will perform either Roux-en-Y or gastric sleeve resection.

SUMMARY:
Obesity is a chronic metabolic condition characterized by excessive accumulation of body fat, which triggers physiological mechanisms that increase the risk of a wide range of health problems. The most effective treatment for severe obesity is metabolic-bariatric surgery, which can lead to a 15-20% weight reduction, significantly lowering the risks of illness and death. However, the success of this surgery can be threatened by poor eating habits after the procedure. The main goal of this study is to enhance the long-term effectiveness of bariatric surgery by combining it with non-invasive brain stimulation (tDCS) targeting inhibitory centers before the operation. Additionally, the investigators aim to comprehensively monitor patients before and after surgery, focusing on investigating changes in brain function associated with the achieved weight loss.

DETAILED DESCRIPTION:
Obesity, defined as a body mass index (BMI) above 30 kg/m² or through other body composition measurements like waist circumference or body fat percentage, is a major risk factor for cardiovascular, neurological, and oncological diseases. It is one of the leading causes of mortality in both men and women. The prevalence of obesity is increasing globally, particularly among younger populations, surpassing undernutrition and posing significant health and socio-economic challenges.

Excess fat accumulation, a hallmark of obesity, impacts the structure and function of nearly all organ systems. This occurs through both physical mechanisms, such as fat deposition around organs, and functional mechanisms, including chronic low-grade inflammation, insulin resistance, dyslipidemia, and altered hormone production and regulation by adipose tissue.

While various therapies have been developed to address the negative effects of obesity on body structure and function, early interventions like lifestyle changes and pharmacotherapy have shown only mild and often temporary weight reduction. These approaches frequently lead to cyclical weight changes, which have been linked to increased cardiovascular risk.

Bariatric surgery has emerged as the most effective treatment for severe obesity, delivering significant and long-lasting weight reduction compared to lifestyle modifications. While lifestyle interventions typically achieve a weight loss of 5-10%, bariatric surgery can result in reductions of 15-20%. However, a notable challenge is the risk of failure, primarily due to noncompliant eating behaviors after surgery. Approximately 40% of individuals with extreme obesity are at high risk of experiencing suboptimal outcomes following bariatric surgery.

To address this issue, our project aims to improve the sustainability of bariatric surgery outcomes by incorporating neuromodulation before the procedure. Specifically, the investigators propose using transcranial direct current stimulation (tDCS) to enhance prefrontal inhibitory control by targeting the left dorsolateral prefrontal cortex (lDLPFC). This home-based, non-invasive brain stimulation method seeks to improve behavioral regulation, potentially reducing the likelihood of postoperative complications related to eating habits.

Additionally, researchers aim to identify neural, cognitive, and behavioral predictors of successful bariatric surgery outcomes. By examining these factors, investigators plan to optimize treatment strategies, ensuring more effective and sustainable results for individuals undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with severe or morbid obesity (determined by BMI > 35 or 40 kg/m2, respectively) eligible for BS treatment in compliance with the current guidelines
* Subjects who meet reduced control over eating behavior (disinhibition) criteria in the Eating Habits Questionnaire

Exclusion Criteria:

* Subjects unable to provide informed consent and those unable to understand and cooperate with study-related procedures (based on the physician's discretion)
* Subjects with a personal history of ischemic heart disease, myocardial infarction, stroke, heart failure, and atrial fibrillation
* Subjects who have already undergone BS treatment in the past
* Pregnant subjects or subjects that plan on becoming pregnant during the study.
* Subjects deemed unsuitable for the study based on expert evaluation (e.g., by a physician or neuropsychologist) will be excluded.
* Subjects with dreadlocks (problematic for the EEG)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive impulse control measured via food-modified Go/No-Go task | Baseline, 1 month and 6 months.
  The cognitive task is used to assess response inhibition, particularly in the context of food-related stimuli. It is a variation of the standard Go/No-Go task, where participants must respond quickly to "Go" stimuli (low-calorie item) while withholding responses to "No-Go" stimuli (high-calorie item). Researchers analyze reaction times, accuracy, and commission errors (responses to No-Go stimuli) to evaluate impulse control.

SECONDARY OUTCOMES:
Brain activation related to cognitive control assessed using a multichannel EEG system | Baseline, 1 month and 6 months.
  The investigators will evaluate brain activity in response to food-modified Go/No-Go stimuli and during rest, using Time-Frequency Analysis, focusing on theta and beta power.
Body bioimpedance analysis measured with the InBody 720 device | Baseline, 1 month and 6 months.
  Patients, wearing light clothing and standing barefoot with their legs slightly apart, will hold the device's sensors. Within seconds, the device calculates parameters such as total body water, fat mass, muscle mass, and segmental composition.
Food craving of patients assessed using Food Craving Questionnaire - Trait | Baseline, 1 month and 6 months.
  The questionnaire has 21 items with a response scale 1-6, higher score means stronger cravings.
Eating habits of patients assessed using the Three-Factor Eating Questionnaire | Baseline, 1 month and 6 months.
  The Questionnaire has 51 items in total, 36 items ask for true/false judgment, and 15 items are scored on a 4-point Likert-type scale, each item scores either 0 or 1 point, the minimum score for factors Cognitive Restraint, Disinhibition, and Hunger is 0-0-0, the possible maximum score is 21-16-14.

CONTACTS AND LOCATIONS:
Overall Officials: Irena Rektorová, Prof., Principal Investigator — Cetral European Institute of Technology
Locations (2):
- Czechia (2):
  - Saint Anne's University Hospital, Brno, Czechia
  - Central European Institute of Technology Masaryk University, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided